CLINICAL TRIAL: NCT03265977
Title: A Randomized, Placebo Controlled, Double-Blind Phase II Study to Evaluate Safety, Immunogenicity, and Prevention of Infection With Mycobacterium Tuberculosis (Mtb) of H56:IC31 in Healthy Adolescents
Brief Title: A Phase II Study of H56:IC31 in Healthy Adolescents
Acronym: A-043
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Design, sponsorship changed prior to initiation. No study procedures done.
Sponsor: Aeras (Other)
Collaborators: Statens Serum Institut (Other); Aurum Institute (Other); South African Tuberculosis Vaccine Initiative (Other); Oslo University Hospital (Other); University of Copenhagen (Other); University of Bergen (Other); National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A-043
Record Dates: First submitted 2017-08-24; First posted 2017-08-29 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Tuberculosis Infection
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled in two cohorts. Within each cohort participants will be randomized in a 1:1 ratio to receive either H56:IC31 (5 ug H56/500 nmol IC31) or placebo intramuscularly (IM) on Days 0 and 56.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Random numbers generated by IWRS; Stratified by site. Syringes are masked with a translucent colored label, in order to maintain the study blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H56:IC31 (Experimental): 5 ug H56/500 nmol IC31, 0.5 mL Intramuscular (IM), Days 0 and 56
  Interventions: Biological: H56:IC31
- Placebo (Placebo Comparator): Normal saline, 0.5 mL IM, Days 0 and 56
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: H56:IC31 — The H56 antigen is a fusion protein created from 3 Mtb antigens: antigen 85B (Ag85B), ESAT-6, and Rv2660c.
  Arms: H56:IC31
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
This clinical trial will evaluate safety, immunogenicity, and efficacy (prevention of Mtb infection as measured by IGRA conversions) of H56:IC31 in remotely BCG vaccinated adolescents.

DETAILED DESCRIPTION:
This clinical trial will evaluate safety, immunogenicity, and prevention of Mtb infection, (measured by IGRA conversion) of H56:IC31 in remotely BCG vaccinated adolescents. A TB vaccination strategy incorporating H56:IC31 in adolescents or young adults, if found to prevent Mtb infection, would likely have a major impact on TB disease, TB transmission, and control of the epidemic. If vaccination with H56:IC31 is shown to prevent infection with Mtb in this proof of concept study in adolescents, additional larger scale studies examining the impact on TB disease in more diverse populations would be warranted.

Primary objectives

* To evaluate the safety profile of H56:IC31 compared to placebo in HIV-uninfected, remotely BCG vaccinated adolescents.
* To evaluate prevention of Mtb infection by H56:IC31 compared to placebo, as measured by rates of conversion using an ESAT-6 free IGRA.

Secondary objectives

* To evaluate prevention of Mtb infection by H56:IC31 compared to placebo, as measured by rates of sustained conversion using an ESAT-6 free IGRA.
* To evaluate trends in ESAT-6 free IGRA prolonged/sustained conversions and late reversions (i.e., through more than 6 months post initial conversion) in ESAT-6 free IGRA converters.
* To investigate the immunogenicity of H56:IC31 in HIV-uninfected, remotely BCG vaccinated adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Has completed the written informed consent and assent process
2. Is age ≥12 years and ≤17 years on Study Day 0
3. Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study
4. For female participants: agrees to avoid pregnancy from 21 days prior to Study Day 0 through 6 months after the last study vaccination. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, or intrauterine device (IUD)
5. Has general good health, confirmed by medical history and physical examination
6. Had BCG vaccination at least 5 years ago documented by confirmation of parent/guardian that the participant received all childhood vaccines or by presence of healed BCG scar
7. Tests ESAT-6 free IGRA and QFT-Plus negative at screening, using a pre-determined threshold for ESAT-6 free IGRA and the manufacturer's recommended threshold for QFT-Plus of 0.35 IU/mL in either of the TB antigen tubes after nil-subtraction

Exclusion Criteria:

1. Acute illness on Study Day 0
2. Axillary temperature ≥37.5 °C on Study Day 0
3. Abnormal laboratory values from the most recent blood collected prior to randomization as follows (abnormal results may be repeated once and if found to be resolved the participant will not be excluded):

   * Laboratory evidence of hematologic disease (white blood cell count <3000/mm^3 or >11,500/mm^3; hemoglobin <0.9 times the lower limit of normal of the testing laboratory, by age and gender; absolute neutrophil count <1300/mm^3; absolute lymphocyte count <1000/mm^3).
   * ALT, AST, alkaline phosphatase, total bilirubin, creatinine, blood urea nitrogen (BUN) >1.25 times the ULN
4. Urinalysis abnormality greater than Grade 1 on the Toxicity Scale (with the exception of hematuria in a menstruating female), or urinalysis abnormality judged clinically significant by the investigator
5. History or evidence of any clinically significant systemic disease, or any acute or chronic illness that might affect the safety, immunogenicity, or efficacy of investigational product in the opinion of the investigator
6. History of treatment for active TB disease or latent Mtb infection
7. History or evidence, including chest X-ray, of active TB disease
8. Shared household with an individual receiving anti-TB treatment, or known to have incompletely treated culture or smear positive TB, at screening
9. History of autoimmune disease or immunosuppression
10. Used immunosuppressive medication within 42 days before Study Day 0 (inhaled and topical corticosteroids are permitted)
11. Received immunoglobulin or blood products within 42 days before Study Day 0
12. Received any investigational drug or investigational vaccine within 180 days before Study Day 0, or planned participation in any other clinical trial during the study period
13. Received investigational TB vaccine at any time prior to Study Day 0
14. Planned administration/administration of a licensed vaccine in the period starting 28 days before and ending 28 days after each dose of investigational product
15. History or laboratory evidence of any past or present possible immunodeficiency state including, but not limited to, any laboratory indication of HIV 1 infection
16. History of allergic disease or reactions, including eczema, likely to be exacerbated by any component of the investigational product
17. History of alcohol or drug abuse
18. Any female currently pregnant or lactating/nursing, or positive urine pregnancy test during screening or Study Day 0
19. Received a tuberculin skin test (TST) within 3 months (90 days) prior to Study Day 0.
20. Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the participant will comply with the protocol.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | Day 0 through month 24
  To evaluate the safety profile of H56:IC31 compared to placebo in HIV-uninfected, previously BCG vaccinated adolescents.
ESAT-6 free IGRA conversion from a negative to positive test at any time point after Day 84 and through end of follow-up for the primary endpoint. | Day 84 through month 24
  To evaluate prevention of Mtb infection by H56:IC31 compared to placebo, as measured by rates of conversion using an ESAT-6 free IGRA.

SECONDARY OUTCOMES:
Primary ESAT-6 free IGRA conversion from a negative to a positive test | Day 84 through month 24
  Primary ESAT-6 free IGRA conversion from a negative to a positive test at any time point after Day 84 and through end of follow up for the primary endpoint, AND persisting without ESAT-6 free IGRA reversion from a positive to a negative test through 6 months after ESAT-6 free IGRA conversion.
Primary ESAT-6 free IGRA conversion from a negative to a positive test | Day 84 through end of study (approximately 24 months)
  Primary ESAT-6 free IGRA conversion from a negative to a positive test at any time point after randomization and through end of follow up for the primary endpoint, AND persisting without ESAT-6 free IGRA reversion from a positive to a negative test through 6 months after ESAT-6 free IGRA conversion.
Initial ESAT-6 free IGRA reversion from a positive to a negative test at any time point after primary ESAT-6 free IGRA conversion through the end of follow up. | Day 84 through month 24
  To evaluate trends in ESAT-6 free IGRA prolonged/sustained conversions and late reversions (i.e., through more than 6 months post initial conversion) in ESAT-6 free IGRA converters.
Percentage of CD4+ and CD8+ T cells that express IFN-γ, TNF, and/or IL-2 alone or in combination in response to stimulation with peptide pools representing the entire amino acid sequence of the vaccine antigens. | Day 0 through month 24
  Immunogenicity of H56:IC31 in HIV-uninfected, previously BCG vaccinated adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Dereck Tait, MD, Study Director — Aeras
Locations (4):
- South Africa (3):
  - Aurum Institute - Klerksdorp, Klerksdorp
  - Aurum Institute - Rustenburg, Rustenburg
  - Aurum Institute - Tembisa, Tembisa
- National Institute for Medical Research, Mwanza, Isamilo Area, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided